CLINICAL TRIAL: NCT06950385
Title: A Phase 3, Multi-Site, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of eRapa to Improve Clinical Outcomes in Patients With Familial Adenomatous Polyposis
Brief Title: Phase 3 Trial of eRapa in Patients With Familial Adenomatous Polyposis
Acronym: SERENTA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rapamycin Holdings Inc. (Industry)
Collaborators: Biodexa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTX230-301
Record Dates: First submitted 2025-04-10; First posted 2025-04-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Familial Adenomatous Polyposis (FAP)
Keywords: FAP; Polyposis; Polyps; ileal pouch
MeSH Terms: conditions — Adenomatous Polyposis Coli; Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- eRapa (Experimental): 0.5 mg eRapa once a day (QD) every other week
  Interventions: Drug: eRapa (encapsulated rapamycin)
- Placebo (Placebo Comparator): Placebo once a day (QD) every other week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eRapa (encapsulated rapamycin) — 0.5 mg capsules for oral use; white opaque capsule filled with off-white powder; Trial intervention will be provided in 28-count round high-density polyethylene bottles with a polypropylene child-resistant screw cap and foil induction seal.
  Arms: eRapa
Drug: Placebo — Capsules in 28-count round high-density polyethylene bottles with a polypropylene child-resistant screw cap and foil induction seal.
  Arms: Placebo

SUMMARY:
The main goal of this clinical trial is to learn if the drug eRapa works to slow down the progression of disease in patients diagnosed with Familial Adenomatous Polyposis (FAP). Researchers will compare eRapa to Placebo. The questions to be answered by this trial are:

* Does taking eRapa help to slow down the progression of the disease in patients with FAP?
* Is eRapa a safe treatment for patients diagnosed with FAP?
* What is the effect of eRapa on the number of polyps found in GI tract of patients diagnosed with FAP?
* How does treatment with eRapa affect a patient's quality of life?

Participants will:

* Take eRapa or placebo once per day every other week until disease progresses (gets worse), stops taking part in the trial or dies.
* Visit the clinic once every 3 months for check ups and tests.
* Have an endoscopy at the start of the trial and then every 6 months to check on whether the disease is getting better or worse.

DETAILED DESCRIPTION:
This is a Phase 3, multi-site, prospective, randomized, double-blind, placebo-controlled trial of eRapa administered to patients with FAP who are at high risk of disease progression. 168 patients with FAP will be enrolled in the trial and randomized 2:1 to receive 0.5 mg eRapa or matching placebo orally, once a day (QD) every other week. There is no minimum treatment duration as this is an event-driven trial; however, the intervention period will continue until disease progression, participant withdrawal from treatment, or until the overall trial endpoint is reached. Participant eligibility is restricted to patients under active surveillance for genetic or clinically diagnosed FAP and who have an intact colon; who are postcolectomy/subtotal colectomy and have documented residual polyps in the rectum/sigmoid or who are post-proctocolectomy with ileal-pouch anal anastomosis and documented polyps in the pouch. Eligible participants will undergo a baseline endoscopy and subsequent endoscopic procedures performed every 6 months to monitor for disease progression.

Randomized patients will be stratified based on the following disease characteristics:

* Intact colon versus post-surgical resection with retained rectum/sigmoid or pouch, and
* Duodenal polyposis (current Spigelman stage score ≤2 versus Spigelman stage score ≥3) For the purposes of this trial, high-risk for disease progression is defined as meeting one of the following:
* Patients who have intact colons and have >100 polyps but ≤500 polyps
* Patients who have retained rectum/sigmoid or ileal-pouch-anal anastomosis and have ≥10 polyps that are ≥3 mm in diameter, or
* Patients who have a history of duodenal polyposis Spigelman stage score of 3 or 4 with at least 1 duodenal polyp that has been removed within 18 months of screening.

Trial assessments should be conducted as per the Schedule of Activities with a visit occurring about once every 3 months.

Assessment of Spigelman stage will not require a biopsy unless the lesion has an abnormal appearance and/or is ≥10 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age inclusive.
2. Participant must have documented FAP, confirmed by adenomatous polyposis coli genotype mutation testing.
3. Participant must have at least 1 of the following high-risk features: >100 polyps but ≤500 polyps in the colon, or ≥10 polyps in the retained rectum/sigmoid or ileal pouch (≥3 mm in size), or Spigelman stage 3 or 4 with at least 1 polyp ≥10 mm to be removed at baseline or on endoscopy performed within 18 months of screening.
4. Contraceptive use by participants or participant partners until at at least 12 weeks after stopping study treatment.
5. Agree not to donate gametes for the purpose of reproduction until at at least 12 weeks after stopping study treatment.
6. Willing to undergo endoscopic evaluation.

Exclusion Criteria:

1. Participant has unresected or incompletely resected high-grade dysplasia or cancer within the duodenum, colon, rectum, or ileal pouch at screening endoscopy.
2. Participant has any polyps ≥8 mm in the duodenum, colon, rectum, or ileal pouch remaining after screening endoscopy (polyps ≥8 mm are to be resected during screening endoscopy).
3. Participant has had surgery within 6 weeks of the trial.
4. Participant has active malignancy or history of malignancy diagnosed within 24 months of first dose of trial intervention.
5. Participant has a history of, or currently has, an acquired or primary (congenital) immunodeficiency.
6. Participant has active and clinically significant tuberculosis (positive Quantiferon Gold test), bacterial, fungal, or viral infection, including human immunodeficiency virus (HIV).
7. Participant has any medical or social condition that, in the opinion of the Investigator, might increase participant risk if enrolled, prevent participant compliance to trial procedures, or present an unacceptable confound to safety or clinical trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in high-risk patients with FAP treated with eRapa versus placebo. | 3 years
  * Death from any cause
  * Cancer/high-grade dysplasia
  * Major FAP-related surgery (e.g., colectomy, proctectomy, total proctocolectomy with ileal pouch anal anastomosis [IPAA], pouch resection, ileostomy, duodenectomy, or surgical ampullectomy)
  * Advancement of Spigelman stage (not related solely to increase in polyp number)
  * Meets criteria for surgery (consistent with United States [US] and European Union [EU] practice guidelines) (Yang, Gurudu et al. 2020, Zaffaroni, Mannucci et al.2024)
  * Retained rectum/sigmoid or pouch (≥10 polyps ≥3 mm in size at baseline)
  * Duodenum (Stage 3/4 and at least 1 polyp ≥10 mm removed in last 18 months)

SECONDARY OUTCOMES:
The safety and tolerability of eRapa in patients with FAP | 3 years
  -Frequency of all grades (as per the Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) treatment-emergent adverse events (TEAEs) in participants receiving eRapa;
  * Frequency of Grade 3 and higher (as per the CTCAE v5.0) TEAEs in participants receiving eRapa
  * Percentage of participants discontinuing eRapa treatment due to adverse drug reactions (ADRs)
The effect of eRapa treatment on GI polyposis in patients with FAP | 3 years
  * Percent change from baseline in the PB (i.e., the sum of the diameters of all polyps >3 mm) at 6, 12, 18, 24, 30, and 36 months as observed by surveillance endoscopy Note: The total PB will be based on polyps observed in the upper GI tract (duodenum) and the lower GI tract (colon, retained rectum/sigmoid or pouch)
  * Percent change from baseline in the PB in the upper GI tract (duodenum) at 6, 12, 18, 24, 30, and 36 months as observed by upper endoscopy
  * Percent change from baseline in the PB in the lower GI tract (colon, retained rectum/ sigmoid or pouch) at 6, 12, 18, 24, 30, and 36 months as observed by lower endoscopy
The effect of eRapa treatment on Spigelman stage score in patients with FAP | 3 years
  Change from baseline in Spigelman stage score at 6, 12, 18, 24, 30, and 36 months
The effect of eRapa treatment on quality-of-life measures, assessed by the 5 level EuroQoL-5 Dimension (EQ-5D-5L) | 3 years
  -Change from baseline in EQ-5D-5L score at 6, 12, 18, 24, 30, and 36 months;
Determine the immunomodulating effect of eRapa treatment in patients with FAP | 3 years
  • Change from baseline in T cell phenotypes and function at 12, 24, and 36 months
The effect of eRapa treatment on quality-of-life measures, assessed by EORTC-30 | 3 years
  -Change from baseline in EORTC-30 score at 6, 12, 18, 24, 30, and 36 months;

CONTACTS AND LOCATIONS:
Overall Officials: Gary Shangold, MD, Study Director — Biodexa
Locations (24):
- United States (16):
  - City of Hope, Arcadia, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Digestive & Liver Center of Florida, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Department of Surgery, Section of Colon Rectal and Surgery, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Washington - Fred Hutchinson, Seattle, Washington
- Copenhagen University Hospital, Copenhagen, Denmark
- Universitätsklinikum Bonn, Bonn, Germany
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Radboud University Medical Center, Nijmegen
- Hospital Oncologico - Puerto Rico Medical Center, Rio Piedras, Puerto Rico
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Comarcal de Inca, Inca
  - Hospital La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided